CLINICAL TRIAL: NCT04458701
Title: Prospective Data Analysis of a Quality Improvement Initiative for Perioperative Hemodynamic Optimization Therapy and Postoperative Outcomes in Patients Undergoing High-Risk Cardiac Surgery
Brief Title: Prospective Data Analysis of a Quality Improvement Initiative in High Risk Cardiac Surgery Patients
Status: Completed | Type: Observational
Sponsor: Loma Linda University (Other)
Collaborators: Edwards Lifesciences (Industry)
Responsible Party: Principal Investigator, Davinder Ramsingh, MD, MD, Loma Linda University
Other Study IDs: 5170287
Record Dates: First submitted 2020-07-01; First posted 2020-07-07 (Actual); Last update posted 2020-08-31 (Actual); Status verified 2020-08

CONDITIONS: Coronary Artery Bypass Graft
MeSH Terms: interventions — Hemodynamic Monitoring

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

INTERVENTIONS:
Device: Hemodynamic monitoring — This is a comprehensive hemodynamic management strategy that would-be initiated in the operating room post-bypass and then continued for the first 12 hours in the intensive care unit

SUMMARY:
This project is designed to assess the impact of implementing a hemodynamic optimization protocol, utilizing flow guided parameters that is provided by technology from Edwards Lifesciences, for patients undergoing high risk cardiac surgery. Importantly, this project is being targeted as a QI initiative because there is no evaluation of new technology or procedures. All technologies and procedures are currently being used for patients undergoing cardiac surgery. Rather this project is evaluating the implementation of a multi-dispclinary developed protocol that seeks to remove variability in which providers are currently treating patients hemodynamics during and acutely after cardiac surgery. Previous research has demonstrated that implementation of hemodynamic management protocols improves perioperative outcome in surgical patients. This project seeks to evaluate the impact of implementing this protocol as the new clinical standard for high-risk cardiac surgery patients. Specifically, this protocol would be a comprehensive hemodynamic management strategy that would-be initiated in the operating room post-bypass and then continued for the first 12 hours in the intensive care unit (see figure below). To restate, all technologies and procedures are currently being performed for these patients, however, there has not been a protocol guiding how practionioners use this technology. The project is evaluating the impact of protocolized treatment strategies. Importantly this protocol has been designed, reviewed and agreed by the motivation of the physicians who are currently responsible for managing these patients hemodynamics. Since this project does involve alterations in procedures or technologies we are seeking to proceed as a quality improvement project. Additionally the protocol is one that has been reviewed and agreed to provide the optimal management strategy for these patients. This again is the overall focus of this project, to implement a hemodynamic management protocol to improve outcomes in patients undergoing cardiac surgery.

ELIGIBILITY:
Inclusion Criteria:

(1) the procedure was a first-start case, (2) the procedure was scheduled, (3) the procedure is considered non-emergent, and (4) the cardiac surgery required cardiopulmonary bypass

Exclusion Criteria:

(1) Patients less than 18 years of age, (2) failure to undergo CPB, (3) non-first-start or emergent classification, (4) as well those who did not receive at least 12 hours of inotropic and/or vasoconstrictive agents were excluded from the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All adult high risk cardiac surgical patients undergoing procedures requiring cardiopulmonary bypass. High risk was defined, a priori, as patients who are expected to require an inotropic and/or vasoconstrictive agent for more than 12 hours post-CPB.
Sampling Method: Non-Probability Sample
Enrollment: 195 (Actual)
Dates: Start 2019-01-17 (Actual); Primary Completion 2020-02-01 (Actual); Study Completion 2020-06-30 (Actual)

PRIMARY OUTCOMES:
Length of Stay | days
  ICU length of stay

SECONDARY OUTCOMES:
Major postoperative complications identified as: | during hospitalization
  1) incidence of stroke, (2) incidence of renal failure (defined as a threefold or greater rise in creatinine or new dialysis requirement), (3) prolonged intubation (>24 hours), and/or (4) a sternal wound infection.
Hospital length of stay | days
30-day readmission | days

CONTACTS AND LOCATIONS:
Overall Officials: Davinder Ramsingh, MD, Principal Investigator — Loma Linda University
Locations (1):
- Loma Linda University Medical Center, Loma Linda, California, United States

IPD SHARING:
Plan to Share IPD: No